CLINICAL TRIAL: NCT04672265
Title: A Randomized Trial to Increase Access to Breast Cancer Screening by Invitation Language Among Immigrants in Norway
Brief Title: Increasing Access to Breast Cancer Screening Among Immigrants
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Paula Berstad, Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19/218; 213396 (Other Grant/Funding Number: The Norwegian Cancer Society)
Record Dates: First submitted 2020-11-16; First posted 2020-12-17 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Cancer Screening
Keywords: cancer screening; breast cancer; non-native; immigrant; participation rate; invitation; information
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are randomized to receive the invitation in the major official native language in the country the participant is born and Norwegian, or in Norwegian only, consecutively when it is their turn to be invited to screening.
Who Masked: Participant
Masking Description: The screening invitees randomized to the control group are not informed about this study. They receive "care as usual", the screening invitation letter in Norwegian language.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mother tongue and Norwegian (Experimental): Written material related to screening sent to the invitee in two languages.
  Interventions: Other: Mother tongue and Norwegian
- Norwegian (No Intervention): Written material related to screening sent to the invitee in Norwegian only.

INTERVENTIONS:
Other: Mother tongue and Norwegian — The screening invitation letter, the information leaflet, the reminder letter and the result letter will be sent in two languages; an official language in the country where the invitee is born, and Norwegian.
  Arms: Mother tongue and Norwegian

SUMMARY:
The investigators aim to test whether inviting immigrants to breast cancer screening with a letter in their mother tongue in addition to the standard letter in Norwegian changes screening uptake in these immigrant groups, compared with a comparable group who receive the invitation in Norwegian only,

DETAILED DESCRIPTION:
Women in selected immigrant groups according to birth country will be invited to screening and randomized in a 1:1 ratio to receive the screening invitation and information material 1) in the major official native language in the country the invitee is born in addition to Norwegian (intervention group), or 2) only Norwegian (control). The 13 selected countries of origin are Poland, the Philippines, Pakistan, Somalia and Arabic speaking countries (Iraq, Syria, Morocco, Lebanon, Algeria, Egypt, Palestine, Sudan and Tunisia). The five intervention languages will thus be Polish, English, Urdu, Somali and Arabic.

ELIGIBILITY:
Inclusion Criteria:

* Invited to screening program during the study recruitment period (January 2021-June 2022)
* The registered country of birth of the invitee is one of the following; Poland, Pakistan, Philippines, Somalia, Iraq, Syria, Morocco, Lebanon, Algeria, Egypt, Palestine, Sudan and Tunisia

Exclusion Criteria:

* Not reached with the screening invitation letter because of wrong address or similar

Ages: 48 Years to 73 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11355 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Screening attendance | 0-6 months after sent screening invitation letter
  Attendance in breast cancer screening programme (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Berstad, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Oslo University Hospital, Cancer Registry, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hofvind S, Iqbal N, Thy JE, Mangerud G, Bhargava S, Zackrisson S, Berstad P. Effect of invitation letter in language of origin on screening attendance: randomised controlled trial in BreastScreen Norway. BMJ. 2023 Sep 19;382:e075465. doi: 10.1136/bmj-2023-075465. PMID 37726122

DOCUMENTS (1):
  • Study Protocol (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT04672265/Prot_000.pdf